CLINICAL TRIAL: NCT05916612
Title: Influence of Right Ventricular Function on Changes in Exercise Capacity After LVAD
Status: Withdrawn | Type: Observational
Why Stopped: Decision not to move forward with study.
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Steven J. Keteyian, Principle Investigator, Henry Ford Health System
Other Study IDs: Sciamanna01
Record Dates: First submitted 2017-08-16; First posted 2023-06-23 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Left Ventricular Assist Device
Keywords: LVAD; Cardiopulmonary stress test; Right ventricular dysfunction; Stage D heart failure
MeSH Terms: conditions — Ventricular Dysfunction, Right

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an exploratory project with the purpose to describe the responses of the right ventricle (RV) and gas exchange during exercise in patients scheduled to undergo left ventricular assist device (LVAD) implant. Such information might be used to predict the likelihood of RV failure after LVAD implant. Additionally, although patients that undergo LVAD implantation have improved quality of life and survival, their exercise tolerance (although improved) remains markedly reduced compared to healthy subjects. No studies have used cardiopulmonary stress testing and echocardiography to assess cardiac function and gas exchange with LVAD implantation to determine potential factors responsible for their limited function. The aims of this study are as follows:

1. To assess the impact of right ventricle (RV) dysfunction on functional capacity before and after left ventricular assist device (LVAD) implant
2. To determine if the combined use of preoperative clinical, CPX and echo data can assist in predicting who will meet target improvements in functional capacity after LVAD implant.

DETAILED DESCRIPTION:
Prior to the 21st century, the management of patients with end stage heart failure with a reduced ejection fraction (HFrEF) was very limited. For optimal candidates only, heart transplantation may be an option. However, donor hearts are a limited resource in which supply is greatly less than demand. For those patients that are either not candidates for transplantation or never received a compatible heart offer, medical therapy was the only option. Unfortunately patients with end stage HFrEF on medical therapy have a 1 year mortality of greater than 50%. Over the past several decades development of durable left ventricular assist devices (LVAD) has given many end stage heart failure patients another therapeutic option. Compared to optimal medical therapy, these devices have demonstrated significant superiority with improved quality of life and survival benefit (Rose et al. NEJM, 2001). Since their development these devices have undergone many modifications to improve outcomes and reduce complications. However, unfortunately since these devices only support a failing left ventricle, their success is dependent on adequate right ventricular function. Therefore, when considering LVAD implantation, it is imperative that thorough RV assessment takes place in order to avoid implanting these devices in patients in which the RV will subsequently fail. Several studies have investigated clinical, laboratory, hemodynamic and resting echo parameters to help determine which patients have right ventricles that may or may not fail after LVAD implantation. Unfortunately no such risk models or parameters are both greatly sensitive and specific. Consequently, anywhere from 10-40% of LVAD implantations are complicated by RV failure (Lampert and Teuteberg. J of Heart and Lung Transplant, 2015). No studies to date have assessed the right ventricle during exercise testing to determine if exercise-induced parameters could help better predict which patients could undergo LVAD implantation not complicated by RV failure.

This is an exploratory project with the purpose to describe the responses of the right ventricle (RV) and gas exchange during exercise in patients scheduled to undergo left ventricular assist device (LVAD) implant. Such information might be used to predict the likelihood of RV failure after LVAD implant. Additionally, although patients that undergo LVAD implantation have improved quality of life and survival, their exercise tolerance (although improved) remains markedly reduced compared to healthy subjects. No studies have used cardiopulmonary stress testing and echocardiography to assess cardiac function and gas exchange with LVAD implantation to determine potential factors responsible for their limited function. The aims of this study are as follows:

1. To assess the impact of right ventricle (RV) dysfunction on functional capacity before and after left ventricular assist device (LVAD) implant
2. To determine if the combined use of preoperative clinical, CPX and echo data can assist in predicting who will meet target improvements in functional capacity after LVAD implant.

The purposes of this pilot study, as described above, would add to the literature by providing initial insights into RV characteristics during rest and stress (exercise) both before and after LVAD implantation. This information may help guide future studies designed to better predict which patients would or would not develop RV failure after LVAD implantation.

ELIGIBILITY:
Inclusion Criteria:

* Stage D heart failure with reduced ejection fraction
* EF <25%
* Eligible for implantation of left ventricular assist device (LVAD) as either destination therapy (DT) or bridge to transplantation (BTT)
* Body mass index (BMI) less than or equal to 40

Exclusion Criteria:

* Prior LVAD implantation
* Pt that underwent cardiopulmonary stress test as LVAD workup, however, did not receive LVAD for any reason

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population that will be studied will be adult end stage heart failure patients (Stage D according to American College of Cardiology/American Heart Association staging system) that have reduced ejections fraction of <25%. These patients must be eligible for LVAD implantation.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Right ventricular function with exercise after LVAD implant | 8-12 weeks after LVAD implant
  Echocardiography derived right ventricular function assessment during cardiopulmonary stress testing will be compared before and after LVAD implant

SECONDARY OUTCOMES:
Right ventricular function and quality of life after LVAD implant | 8-12 weeks after LVAD implant
  Correlation of right ventricular function with exercise and quality of life both before and after LVAD implant
Correlation of right ventricular function and functional capacity after LVAD implantation | 8-12 weeks after LVAD implant
  Correlation of right ventricular function before and after LVAD implant assessed by cardiopulmonary stress testing and 6 minute walk test.